CLINICAL TRIAL: NCT05836181
Title: The Effect of Eye Movement Desensitization and Reprocessing Reducing Anxiety, Depressive Symptoms, Blood Pressure, and Heart Rate Variability in Primary Hypertension： A Randomized Controlled Clinical Trial
Brief Title: The Effect of Eye Movement Desensitization and Reprocessing Intervention in Hypertension Patient.
Acronym: EMDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miao-Yi Chen (Other)
Responsible Party: Sponsor-Investigator, Miao-Yi Chen, National Defense Medical Center Student, National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TSGHNDMC
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Eye Movement Desensitization and Reprocessing Intervention; Blood Pressure; Heart Rate Variability; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Movement Desensitization and Reprocessing intervention (Experimental): The goal of EMDR is to help manage physical and mental unpleasant experiences due to hypertension. The intervention group received EMDR therapy included eight phases, each lasting 60-90 minutes, and the intervention consisted of four weekly. In this study, a Nurse practitioner trained in EMDR performs an intervention in an outpatient clinic's quiet, empty room.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing
- Eye Movement Desensitization and Reprocessing control (No Intervention): The control group received routine care and treatment as usual. They did not receive EMDR intervention or counseling.

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing — Effects of Eye Movement Desensitization and Reprocessing on Anxiety, Depression, Quality of Life, Blood Pressure and Heart Rate Variability in Patients with Hypertension.
  Arms: Eye Movement Desensitization and Reprocessing intervention

SUMMARY:
Eye Movement Desensitization and Reprocessing intervention may improve anxiety, depression, systolic blood pressure and heart rate variability in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. age of 20-80 years,
2. diagnosed with primary hypertension as in SBP ≥130 mmHg or DBP ≥80 mmHg,
3. and able to read and understand Chinese or Taiwanese and willing to participate in this study,

Exclusion Criteria:

1. . Secondary hypertension
2. . Hypertension Crisis.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Anxiety | Six month
  HADS-A score
depression symptoms | Six month
  CESD Scale

SECONDARY OUTCOMES:
Blood pressure | Six month
  Blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Chen, miao-yi, Taipei, Neihu, Taiwan

IPD SHARING:
Plan to Share IPD: No